CLINICAL TRIAL: NCT03060096
Title: Stepped-Care Telehealth for Distress in Cancer Survivors
Acronym: Telehealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00047561; 1R21CA198237 (NIH); 5R21CA198237-02 (NIH); 3UG1CA189824-04S1 (NIH); WF-30917CD (Other: NCI); NCI-2017-01840 (Registry Identifier: NCI CTRP); NCT03190291 (obsolete NCT alias)
Record Dates: First submitted 2017-01-31; First posted 2017-02-23 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Anxiety; Depressive Symptoms; Sleep Disturbance; Recurrent Disease; Fatigue; Quality of Life; Cancer
MeSH Terms: conditions — Anxiety Disorders; Depression; Parasomnias; Recurrence; Fatigue; Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by baseline score ≥15 on the GAD-7 and/or on the PHQ-9, indicating severe significant anxiety or depressive symptom. Participants with moderate symptoms only (10-14 on the PHQ-9 and/or 8-14 on the GAD-7) will be block randomized to either the low-intensity stepped care or to the enhanced usual care (EUC control). Participants with moderate to severe symptoms will be block randomized to either the high-intensity stepped care intervention or the EUC control. Block sizes will be chosen randomly to ensure that future assignments cannot be inferred from previous ones.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate Anxiety/depression: Low Intensity Stepped care (Experimental): participants with moderate symptoms (PHQ-9-14; GAD-7: 10-14) will be randomized to either low-intensity stepped care or enhanced usual care. Stepped care consist of a self-guided cognitive behavioral therapy (CBT) workbook to reduce anxiety and depressive symptoms and biweekly (every two weeks) check-in calls from research staff to assess changes in symptom severity/immediate need for psychiatric treatment and provide minimal support.
  Interventions: Other: Moderate Anxiety/depression: Low Intensity Stepped care
- Severe Anxiety/depression: High Intensity Stepped Care (Experimental): Participants with severe symptoms (PHQ-9: 15-27; GAD-7: 15-21) will be randomized to high intensity stepped care (consist of a CBT workbook with accompanying psychotherapy by a Master's-level therapist delivered by telephone) or EUC. EUC consist of information about referrals/resources locally and nationally.
  Interventions: Other: Severe Anxiety/depression: High Intensity Stepped Care
- Enhanced Usual Care Control (EUC) (Active Comparator): Participants randomized to EUC will receive information about local referrals/resources (support groups, mental health providers, etc.). They will also be provided "Facing Forward: Life after Cancer Treatment," a book developed by the NCI to assist with transition from active treatment to survivorship. Participants will receive information on self-help workbooks for anxiety & depressive symptoms. EUC control will receive a copy of the CBT workbook on completion of the study.
  Interventions: Other: Enhanced Usual Care Control

INTERVENTIONS:
Other: Severe Anxiety/depression: High Intensity Stepped Care — The stepped-care Telehealth high intensity intervention is tailored to participants with severe anxiety and depression. Ppts randomized to this group will have 12 weekly psychotherapy sessions delivered by phone with a licensed therapist. Participants will also receive a CBT (cognitive behavioral therapy) workbook including daily exercises to supplement understanding.
  Arms: Severe Anxiety/depression: High Intensity Stepped Care
Other: Moderate Anxiety/depression: Low Intensity Stepped care — The stepped care Telehealth low intensity intervention is tailored to participants with moderate anxiety and depression. Ppts randomized to this group will receive a self-guided CBT workbook and biweekly (every 2 weeks) check-in calls from a research staff person to assess changes in symptom severity and need for treatment/support.
  Arms: Moderate Anxiety/depression: Low Intensity Stepped care
Other: Enhanced Usual Care Control — Participants with moderate to severe anxiety/depression that are randomized to Enhanced Usual Care Control (EUC) will receive information about referrals/resources in their local area (support groups, mental health providers), NCI materials (Facing Forward: Life after Cancer Treatment", self-help workbooks, copy of the CBT (cognitive behavioral therapy) workbook on completion of the study.
  Arms: Enhanced Usual Care Control (EUC)

SUMMARY:
Mental health issues in post-treatment adult cancer survivors are associated with multiple adverse outcomes and may represent a cancer health disparity for rural survivors. The purpose of this study is to test a stepped-care approach tailored to symptom severity based on recent American Society of Clinical Oncology guidelines for reducing emotional distress (anxiety and/or depressive symptoms) and improving secondary outcomes (sleep disturbance, fatigue, fear of recurrence, quality of life) in rural, post-treatment cancer survivors in community oncology settings and to examine intervention costs. The resultant intervention will have great potential for widespread dissemination since it will be manualized, delivered by telephone, and comprised of modules to allow customized treatments for individuals with different cancer types.

DETAILED DESCRIPTION:
Noting the need for evidence-based cancer survivorship care, the American Society of Clinical Oncology (ASCO) published guidelines for screening, assessment, and care of psychosocial distress (anxiety, depression) in adults with cancer. These guidelines recommend screening all adults with cancer for distress and treating those with moderate or severe symptoms using a stepped-care approach tailored to distress severity. While these guidelines apply to survivors with all cancer types across the cancer treatment and survivorship continuum, we have chosen to focus on survivors with non-metastatic breast, colorectal, prostate, uterine, and cervical cancers , as well as those with any stage lymphoma (Hodgkin's or non-Hodgkin's). Further, we have focused on the post-treatment survivorship period 6 months-5 years post-treatment because distress may be more likely to be assessed and addressed after treatment completion. A significant minority of post-treatment survivors is at risk for anxiety and depression symptoms during the five years following the end of treatment and accessible interventions are needed to treat them.

The purpose of this study is to test a method of implementing this stepped-care approach in community oncology practices caring for cancer survivors, using self-directed and stepped-care telehealth approaches based on cognitive-behavioral theory. Our approach is based on a previous trial of telephone-based cognitive behavioral therapy for rural older adults with Generalized Anxiety Disorder (NIMH 1R01MH083664: The Tranquil Moments Study; PI: Brenes), which has demonstrated high acceptability and efficacy for reducing anxiety, worry, and depressive symptoms in a rural geriatric population. This protocol adapts the methods of the previous trial to bring psychosocial care to underserved cancer survivors, many of whom have minimal or no access to mental health providers. Cancer survivors will be recruited through multiple NCI Community Oncology Research Program (NCORP) sites through the NCI-funded Wake Forest NCORP Research Base (WF NCORP RB).

We will obtain data on feasibility, outcome variability, and efficacy for designing a subsequent fully powered randomized controlled trial (RCT) assessing the effects of the intervention on distress in cancer survivors. In the planned larger study, we anticipate that this intervention will: (a) reduce treatment barriers for post-treatment cancer survivors; (b) enhance availability of psychosocial treatment (through use of telephone sessions and a workbook); and (c) result in reductions in anxiety and depressive symptoms in cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Score ≥10 on the GAD-7 and/or a score ≥8 on the PHQ-9, indicating clinically significant anxiety or depressive symptoms, respectively.
* Past history of treated Stage I, II, or III (newly diagnosed or recurrent) breast, colorectal, prostate, gynecologic (to include uterine and cervical) cancers and non-Hodgkin's lymphoma.
* 6-60 months post-treatment (surgery, chemotherapy, and/or radiation therapy) for cancer. Time frame applies to most recent completion of treatment if participant had a cancer recurrence. It is acceptable to be on maintenance or hormonal therapies.
* Participant resides in California, Georgia, Illinois, Kansas, Michigan, Minnesota, Missouri, New Mexico, North Carolina, North Dakota, South Carolina, Virginia, Tennessee, or Wisconsin
* Study-trained therapist in the state where the participant resides.
* Must be able to speak and understand English.
* Must have access to a telephone

Exclusion Criteria:

* Current psychotherapy [regular appointment(s) with a psychologist, counselor, or therapist within the last 30 days prior to randomization].
* Self-reported active alcohol or substance abuse within the last 30 days.
* Past history of prostate cancer or non-Hodgkin's lymphoma with only active surveillance (i.e., no surgery, chemotherapy, or radiation therapy).
* Diagnosis of a second malignancy (except for non-melanoma skin cancers) after a previous diagnosis of breast, colorectal, gynecologic cancers and non-Hodgkin's lymphoma
* Progressive cancer (must be considered no evidence of disease or stable)
* Self -reported history of a diagnosis of dementia from a healthcare provider.
* Self -reported psychotic symptoms in the last 30 days prior to randomization
* Active suicidal ideation (currently reported suicidal plan and intent).
* Any change in psychotropic medications within the last 30 days.
* Hearing loss that would preclude participating in telephone sessions (determined by brief hearing assessment administered by research staff)
* Failure/inability/unwillingness to provide names and contact information for two family members or friends to serve as emergency contacts during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (166):
- United States (166):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - Kaiser Permanente-Fresno, Fresno, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Augusta University Medical Center, Augusta, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Sanford Thief River Falls Medical Center, Thief River Falls, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Sanford Cancer Center Worthington, Worthington, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - AdventHealth Infusion Center Asheville, Asheville, North Carolina
  - AdventHealth Infusion Center Haywood, Clyde, North Carolina
  - AdventHealth Hendersonville, Hendersonville, North Carolina
  - AdventHealth Infusion Center Weaverville, Weaverville, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford South University Medical Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Self Regional Healthcare, Greenwood, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Spartanburg Medical Center - Mary Black Campus, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Bristol Regional Medical Center, Bristol, Tennessee
  - Wellmont Medical Associates Oncology and Hematology-Johnson City, Johnson City, Tennessee
  - Regional Cancer Center at Indian Path Community Hospital, Kingsport, Tennessee
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Wellmont Medical Associates-Bristol, Bristol, Virginia
  - Sovah Health Martinsville, Martinsville, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - VCU Community Memorial Health Center, South Hill, Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Aspirus Medford Hospital, Medford, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Started | 19 | 15 | 34
Completed | 16 | 12 | 32
Not Completed | 3 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC) | Total
Number analyzed (Participants) | 19 | 15 | 34 | 68
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 21 | 38
  >=65 years | 11 | 6 | 13 | 30
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 82] | 63 [40 to 77] | 62 [45 to 78] | 64 [36 to 82]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 18 | 14 | 31 | 63
  Male | 1 | 1 | 2 | 4
  Other | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 3 | 5
  White | 16 | 14 | 30 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 15 | 34 | 68
Generalized Anxiety Disorder (GAD)-7 Score for Anxiety [Mean (Standard Deviation); unit: units on a scale] — The GAD-7 is a self-report measure of symptoms of GAD. Participants rate 7 questions on a scale of 0 (not at all) to 3 (nearly every day); one additional question assesses the interference of these symptoms with functioning. The first 7 questions are summed to create a total score ranging from 0 to 21. Higher scores reflect greater anxiety severity. Scores above 10 are considered to be in the clinical range.
  units on a scale | 8.5 (2.7) | 15.9 (3.8) | 11.4 (5.1) | 11.6 (5.0)
Patient Health Questionnaire (PHQ)-9 Score for Depression [Mean (Standard Deviation); unit: units on a scale] — The possible range is 0-27. A larger score represents more severe depression level.
  units on a scale | 10.5 (3.3) | 17.4 (3.2) | 11.8 (3.7) | 12.7 (4.3)
Insomnia Severity Index (ISI) [Mean (Standard Deviation); unit: units on a scale] — The Insomnia Severity Index (ISI) is 7-item self-report measure of type and severity of insomnia symptoms. Each of the seven items is scored on a 5-point scale, ranging from 0 (lowest) to 4 (highest). The sum of the scores for all seven items yields a total score, which falls within a range of 0 to 28. A higher score indicates a greater level of sleep impairment.
  units on a scale | 14.0 (4.5) | 18.6 (7.2) | 13.8 (6.3) | 14.9 (6.3)
PROMIS Fatigue t-Score [Mean (Standard Deviation); unit: t-score] — PROMIS Fatigue Short Form 8a is a measure of the experience of fatigue and the impact of fatigue on activities across multiple domains. There are eight items rated on a scale of 1(never) to 5 (always) based on how often fatigue was experienced over the last 7 days. The sum of these eight items ranges from a minimum of 8 to a maximum of 40, with higher scores representing more fatigue. This total score is then converted into a t-score based on the PROMIS 8a adult conversion table. The smallest t score is 33.1 and the largest t score is 77.8. A higher t score indicates greater fatigue.
  t-score | 59.0 (6.3) | 64.8 (7.9) | 62.2 (8.4) | 61.9 (7.9)
Fear of Recurrence Inventory Severity Subscale [Mean (Standard Deviation); unit: units on a scale] — The Fear of Cancer Recurrence Inventory (FCRI; severity subscale) will be used to measure self-reported fear of recurrence. This 9-item subscale measures the presence and severity of the intrusive thoughts or images associated with the fear of cancer recurrence. Range is 0 to 36 with higher values representing higher fear of recurrence.
  units on a scale | 21.4 (8.8) | 24.3 (6.4) | 22.8 (7.9) | 22.7 (7.8)
Health Status Questionnaire (SF-36) [Mean (Standard Deviation); unit: units on a scale] — SF-36 consists of 36 items and is organized into eight subscales. Each subscale score is then translated into a linear scale that spans from 0 to 100. A higher score means enhanced quality of life. Two domains as mental health component and physical health component are the results of linear aggregation from the 8 subscales and transforming into T score metric. In this metric, the t score has a mean of 50 and a standard deviation of 10 based on the characteristics of U.S. general population. A higher T-score corresponds to a higher quality of life.
  units on a scale
    Physical Health | 40.9 (10.5) | 38.6 (10.4) | 39.1 (10.1) | 39.5 (10.2)
    Mental Health | 37.4 (10.4) | 28.6 (8.3) | 36.1 (11.3) | 34.9 (10.9)
Impact of Events Scale-Revised (IES-R) Total Score [Mean (Standard Deviation); unit: units on a scale] — The Impact of Events Scale - Revised (IES-R) is a 22-item self-report measure of cancer related distress. The IES-R assesses the frequency with which respondents experience intrusive thoughts, avoidant behaviors, and autonomic arousal specific to one's thoughts and feelings about cancer over the past week. IES- R total score is the sum of the means of the three subscale scores. IES- R total score ranges from 0 to 12. The higher scores indicate higher cancer distress.
  units on a scale | 4.0 (2.1) | 5.4 (2.6) | 4.2 (2.4) | 4.4 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Study Intervention Measured by Retention
Description: Study retention will be estimated by the number of participants who complete the Week 7 and 13 visits
Time Frame: Randomization through completion of study at week 13
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
Participants | 16 | 12 | 32
Statistical Analysis 1: Comparison: Moderate Anxiety/Depression: Low Intensity Stepped Care vs Severe Anxiety/Depression: High Intensity Stepped Care vs Enhanced Usual Care Control (EUC); Test type: Superiority; p = 0.29, Fisher Exact

2. Primary Outcome: Feasibility of Study Intervention Measured by Adherence to Intervention
Description: Intervention adherence will be estimated as the mean proportion of therapy (high-intensity intervention) or check-in (low-intensity intervention) sessions each participant completes.
Time Frame: Randomization through completion of study at week 13
Population: Adherence will be documented as the percentage of therapy sessions completed by each participant in the high intensity intervention group, or the percentage of check-in calls completed within the low intensity intervention group. Since the EUC involved no intervention, there was no data collected to assess adherence for this arm.
Measure: Mean (Standard Deviation); unit: proportion of completed intervention
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 0
proportion of completed intervention | 0.82 (0.34) | 0.78 (0.37) |
Statistical Analysis 1: Comparison: Moderate Anxiety/Depression: Low Intensity Stepped Care vs Severe Anxiety/Depression: High Intensity Stepped Care; Test type: Superiority; p = 0.8, t-test, 2 sided

3. Primary Outcome: Feasibility of Study Intervention Measured by Recruitment Rate
Description: Recruitment rate will be determined by the number of eligible participants who met all eligibility criteria and percent who agreed to participate.
Time Frame: Screening through end of study at week 13
Population: All eligible people that were approached to enroll to this trial.
Measure: Count of Participants; unit: Participants
Groups:
- Recruitment Rate of Entire Study: This is simply looking at the rate of people enrolled that were found to be eligible PRIOR to study entry. This is before randomization into a study group.
Arm/Group | Recruitment Rate of Entire Study
Number analyzed (Participants) | 89
Participants | 68
Statistical Analysis 1: Comparison: Recruitment Rate of Entire Study; Test type: Other; Rate = 0.7640, 95% CI 1-sided [lower limit 0.6783]

4. Primary Outcome: Feasibility of Study Intervention Measured by Accrual Rate
Description: The accrual rate is determined by dividing the overall number of participants recruited in each arm by the total span of 38 months between the start of the first screening for enrollment and the time the study closed to accrual.
Time Frame: Start of study screening time to end of study accrual
Population: All those enrolled.
Measure: Number; unit: participants per month
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
participants per month | 0.5 | 0.4 | 0.9

5. Secondary Outcome: Longitudinal Changes in the Generalized Anxiety Disorder (GAD)-7 Score for Anxiety From Baseline to 13 Weeks
Description: The Generalized Anxiety Disorder (GAD) -7 is a self-report measure of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) symptoms of Generalized Anxiety Disorder (GAD). Longitudinal changes in the GAD-7 will be measured in participants to evaluate the effectiveness of the intervention in reducing anxiety. Patients select 1 of 4 numbers with "0" indicating not all, to "3" indicating nearly everyday. The first 7 questions are summed to create a total score ranging from 0 to 21. Higher scores reflect greater anxiety severity. Scores above 10 are considered to be in the clinical range. GAD-7 scores of 5, 10, 15, and 20 represented mild, moderate, moderately severe, and severe anxiety, respectively.
Time Frame: Screening or baseline (if >30 days since screening), Week 13
Population: Intent to treat analysis of all those participants that completed GAD-7 at baseline and at week 13.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 16 | 12 | 34
score on a scale | -1.1 [-3.8 to 1.5] | -8.6 [-11.4 to -5.7] | -4.1 [-6.3 to -1.8]

6. Secondary Outcome: Longitudinal Changes in the Patient Health Questionnaire (PHQ-9) Score for Depression From Baseline to 13 Weeks
Description: The PHQ-9 is a self-report measure of DSM-IV symptoms of Major Depressive Disorder where participants rate how often they experienced 9 symptoms over past 2 weeks. Patients select 1 of 4 numbers with "0" indicating not all, to "3" indicating nearly everyday. Longitudinal changes in the PHQ-9 will be measured in participants to evaluate the effectiveness of the intervention in reducing depression. The possible range is 0-27. A larger score represents more severe depression level.
Time Frame: Screening or baseline (if >30 days since screening), Week 13
Population: Intent to treat of all participants who have outcome at baseline and 13 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Moderate Anxiety/Depression: Low Intensity: GAD-7: 10-14) will be randomized to either low-intensity stepped care or enhanced usual care. Stepped care consist of a self-guided cognitive behavioral therapy (CBT) workbook to reduce anxiety and depressive symptoms and biweekly (every two weeks) check-in calls from research staff to assess changes in symptom severity/immediate need for psychiatric treatment and provide minimal support.
  Moderate Anxiety/depression: Low Intensity Stepped care: The stepped care Telehealth low intensity intervention is tailored to participants with moderate anxiety and depression. Ppts randomized to this group will receive a self-guided CBT workbook and biweekly (every 2 weeks) check-in calls from a research staff person to assess changes in symptom severity and need for treatment/support.
- Severe Anxiety/Depression: High Intensity: Participants with severe symptoms (PHQ-9: 15-27; GAD-7: 15-21) will be randomized to high intensity stepped care (consist of a CBT workbook with accompanying psychotherapy by a Master's-level therapist delivered by telephone) or EUC. EUC consist of information about referrals/resources locally and nationally.
  Severe Anxiety/depression: High Intensity Stepped Care: The stepped-care Telehealth high intensity intervention is tailored to participants with severe anxiety and depression. Ppts randomized to this group will have 12 weekly psychotherapy sessions delivered by phone with a licensed therapist. Participants will also receive a CBT (cognitive behavioral therapy) workbook including daily exercises to supplement understanding.
Arm/Group | Moderate Anxiety/Depression: Low Intensity | Severe Anxiety/Depression: High Intensity | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
score on a scale | -2.0 [-4.2 to 0.4] | -8.8 [-11.3 to -6.3] | -3.2 [-5.1 to -1.2]

7. Secondary Outcome: Number of Participants With Moderate of Severe Depression (PHQ-9) or Anxiety (GAD-7) at 13 Weeks
Description: A combined variable will be created that indicates if a participant had moderate/severe depression or anxiety at mid- or post-intervention. This is defined as either PHQ-9 or GAD-7 greater than or equal to 15.
Time Frame: Week 13
Population: Intent to treat population of all those with data available at 13 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
Participants | 0 | 2 | 5

8. Secondary Outcome: Longitudinal Changes in the Insomnia Severity Index (ISI) From Baseline to 13 Weeks.
Description: Measure Description: The Insomnia Severity Index (ISI) is 7-item self-report measure of type and severity of insomnia symptoms, including problems with sleep onset, sleep maintenance, or early morning awakening; satisfaction with current sleep pattern; interference with daily functioning; noticing impairment attributed to sleep problems; and level of concern or distress caused by the sleep problem. Each of the seven items is scored on a 5-point scale, ranging from 0 (lowest) to 4 (highest). The sum of the scores for all seven items yields a total score, which falls within a range of 0 to 28. A higher score indicates a greater level of sleep impairment.
Time Frame: Baseline (Week 0), Week 13
Population: Intent to treat population of all with available ISI data at baseline and 13 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
score on a scale | -3.1 [-6.9 to 0.6] | -7.7 [-11.8 to -3.7] | -2.9 [-6.1 to 0.3]

9. Secondary Outcome: Longitudinal Changes in the PROMIS Fatigue Scale From Baseline to 13 Weeks
Description: The Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 8a is a measure of the experience of fatigue and the impact of fatigue on activities across multiple domains. There are eight items rated on a scale of 1(never) to 5 (always) based on how often fatigue was experienced over the last 7 days. The sum of these eight items ranges from a minimum of 8 to a maximum of 40, with higher scores representing more fatigue. This total score is then converted into a t-score based on the PROMIS 8a adult conversion table. The smallest t score is 33.1 and the largest t score is 77.8. A higher t score indicates greater fatigue.
Time Frame: Baseline (Week 0), Week 13
Population: intent to treat population of all those with PROMIS data at baseline and 13 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: t-score
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
t-score | 0.1 [-5.0 to 5.2] | -5.6 [-11.1 to -0.1] | -3.1 [-7.4 to 1.3]

10. Secondary Outcome: Longitudinal Changes in the Fear of Recurrence Inventory Severity Subscale From Baseline to 13 Weeks
Description: The Fear of Cancer Recurrence Inventory (FCRI; severity subscale) will be used to measure self-reported fear of recurrence. This 9-item subscale measures the presence and severity of the intrusive thoughts or images associated with the fear of cancer recurrence. Range is 0 to 36 with higher values representing higher fear of recurrence.
Time Frame: Baseline (Week 0), Week 13
Population: all participants that have FCRI measured at baseline and 13 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate Anxiety/Depression: Low Intensity | Severe Anxiety/Depression: High Intensity | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
score on a scale | -1.7 [-6.3 to 2.9] | -4.7 [-9.6 to 0.3] | -3.1 [-7.0 to 0.8]

11. Secondary Outcome: Longitudinal Changes in the Health Status Questionnaire (SF-36) From Baseline to 13 Weeks
Description: The Health Status Questionnaire (SF-36) functions as a self-reporting tool designed to evaluate an individual's quality of life. It consists of 36 items and is organized into eight subscales. Each subscale score is then translated into a linear scale that spans from 0 to 100. A higher score means enhanced quality of life. Additionally, the questionnaire incorporates two domains as mental health component and physical health component. These domains are the results of linear aggregation from the 8 subscales and transforming into T score metric. In these metrics, the t score has a mean of 50 and a standard deviation of 10 based on the characteristics of U.S. general population for both mental and physical health sub scores. A higher T-score corresponds to a higher quality of life for that subscale.
Time Frame: Baseline (Week 0), Week 13
Population: all participants with recorded SF-36 data at baseline and 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: t-score
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
t-score
  Mental health | 3.4 [-3.0 to 9.7] | 12.2 [5.1 to 19.2] | 4.7 [-0.7 to 10.1]
  Physical health | -1.1 [-7.3 to 5.2] | 1.2 [-5.7 to 8.1] | 0.7 [-4.6 to 6.0]

12. Secondary Outcome: Longitudinal Changes in the Impact of Events Scale-Revised (IES-R) From Baseline to 13 Weeks
Description: The Impact of Events Scale - Revised (IES-R) is a 22-item self-report measure of cancer related distress. The IES-R assesses the frequency with which respondents experience intrusive thoughts, avoidant behaviors, and autonomic arousal specific to one's thoughts and feelings about cancer over the past week. Each item is rated on a 5-point scale ranging from 0("not at all") to 4("extremely"). The higher grade indicates greater stress. IES- R total score is the sum of the means of the three subscale scores. IES- R total score ranges from 0 to 12. The higher scores indicate higher cancer distress.
Time Frame: Baseline (Week 0), Week 13
Population: all participants with IES-R data at baseline and 13 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Moderate Anxiety/Depression: Low Intensity | Severe Anxiety/Depression: High Intensity | Enhanced Usual Care Control (EUC)
Number analyzed (Participants) | 19 | 15 | 34
score on a scale | -0.3 [-1.7 to 1.0] | -1.8 [-3.2 to -0.4] | -0.6 [-1.7 to 0.49]

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Moderate Anxiety/Depression: Low Intensity Stepped Care | Severe Anxiety/Depression: High Intensity Stepped Care | Enhanced Usual Care Control (EUC)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/34
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/15 | 2/34
Other Adverse Events (participants affected / at risk) | 3/19 | 2/15 | 5/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Anxiety/Depression: Low Intensity Stepped Care (N=19) | Severe Anxiety/Depression: High Intensity Stepped Care (N=15) | Enhanced Usual Care Control (EUC) (N=34)
SAE (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Hospitalization/Planned Hip Replacement 1 Day Hospitalization
SAE (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalization/vascular disorder-other; aortic aneurysm
SAE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) — Hospitalization/Acute pyelonephritis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moderate Anxiety/Depression: Low Intensity Stepped Care (N=19) | Severe Anxiety/Depression: High Intensity Stepped Care (N=15) | Enhanced Usual Care Control (EUC) (N=34)
Worsening Anxiety (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) — Worsening Anxiety
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 5 (5) — Depression
Suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) — Suicidal ideation
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Shoulder pain
Diarrhea on and off (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Diarrhea on and off

LIMITATIONS AND CAVEATS:
The study didn't reach the recruitment goal due to slow accrual rates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03060096/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03060096/ICF_001.pdf